CLINICAL TRIAL: NCT02633761
Title: Mifepristone and Misoprostol Versus Misoprostol Alone for Treatment of Fetal Death at 14-28 Weeks of Pregnancy: A Randomized, Placebo-controlled Double-blinded Trial
Brief Title: Mifepristone-misoprostol vs. Misoprostol Alone for Second Trimester Fetal Death
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1019
Record Dates: First submitted 2015-12-08; First posted 2015-12-17 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-01

CONDITIONS: Fetal Death
Keywords: Fetal death; mifepristone; misoprostol
MeSH Terms: conditions — Fetal Death | interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): 200mg mifepristone followed in 24 hours by repeated doses of 200mcg buccal misoprostol given every 3 hours
  Interventions: Drug: Mifepristone; Drug: Misoprostol 200mcg
- Group 2 (Placebo Comparator): placebo followed in 24 hours by 200mcg buccal misoprostol given every three hours.
  Interventions: Drug: Placebo; Drug: Misoprostol 200mcg

INTERVENTIONS:
Drug: Mifepristone — 200mg mifepristone followed in 24 hours by 200mcg buccal misoprostol every 3 hours.
  Arms: Group 1
Drug: Placebo — placebo followed in 24 hours by 200mcg buccal misoprostol every 3 hours.
  Arms: Group 2
Drug: Misoprostol 200mcg — Buccal misoprostol 200mcg

SUMMARY:
The primary aim of this trial is to compare the efficacy of mifepristone-misoprostol versus misoprostol alone for treatment of intrauterine fetal demise between 14 and 28 weeks LMP.

DETAILED DESCRIPTION:
The primary aim of this trial is to compare the efficacy of mifepristone-misoprostol versus misoprostol alone for treatment of intrauterine fetal demise between 14 and 28 weeks LMP. This will be a randomized controlled double-blinded trial of 150 women comparing misoprostol alone to mifepristone plus misoprostol for evacuation of the uterus after fetal demise in the second and third trimester. All women in the trial will undergo routine screening and pre-medical induction care per standard practice at the hospital.

All eligible women agreeing to participate in the study will be randomized to receive one of the following regimens:

1. STUDY GROUP ONE: 200mg mifepristone followed in 24 hours by repeated doses of 200mcg buccal misoprostol given every 3 hours;
2. STUDY GROUP TWO: placebo followed in 24 hours by 200mcg buccal misoprostol given every three hours.

ELIGIBILITY:
Inclusion Criteria:

* Demised fetus of between 14 to 28 weeks duration confirmed by ultrasound
* Have no contraindications to study procedure, according to provider
* Be able to consent to procedure, either by reading consent document or by having consent document read to her
* Be willing to follow study procedures.

Exclusion Criteria:

* Allergies or other contraindications to the use of mifepristone or misoprostol;
* Placental abruption with active hemorrhage,
* Complete placenta previa, extreme uterine structural anomalies, or other contradictions to vaginal delivery of the fetus;
* Presentation in active labor (moderate to severe contractions every 10 minutes or less);
* Transmural uterine scars;
* Four or more previous deliveries.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-04-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Complete uterine evacuation of the fetus and placenta without surgical intervention | 48 hours
  Complete uterine evacuation of fetus and placenta using study drug alone without recourse to any additional surgical intervention

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Bracken, PhD, Principal Investigator — Gynuity Health Projects
Locations (3):
- Mexico (2):
  - Hospital General "Enrique Cabrera", Mexico City
  - National Institute of Perinatology (INPer), Mexico City
- National Ob-Gyn Hospital, Hanoi, Vietnam